CLINICAL TRIAL: NCT04763031
Title: A Pilot Study of Patients With Recurrent Glioblastoma Treated With Maximal Safe Neurosurgical Resection, Intra-Operative Radiation Therapy (IORT) Using the Xoft® Axxent® Electronic Brachytherapy System
Brief Title: Recurrent GBM With Maximal Neurosurgical Removal and Treatment With IORT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No potential patients enrolled since first enrollment on 06/27/2022.
Sponsor: Parkridge Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PMC-3422401
Record Dates: First submitted 2021-02-04; First posted 2021-02-21 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Glioblastoma; GBM; Recurrent GBM
Keywords: Glioblastoma; GBM; Recurrent GBM; Recurrent Glioblastoma; IORT; Intra-Operative Radiation Therapy
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Intervention Model Description: Single 20 Gy (gray) dose of electronic brachytherapy (IORT)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Intra-operative Radiation Therapy - IORT (Experimental): Intra-operative Radiation Therapy - IORT
  Interventions: Radiation: Intra-operative Radiation Therapy - IORT

INTERVENTIONS:
Radiation: Intra-operative Radiation Therapy - IORT — Single dose of 20 Gy
  Other Names: Electronic Brachytherapy

SUMMARY:
The purpose of this study is to assess the safety and efficacy of the Xoft Axxent eBx System when used for single-fraction IORT for recurrent Glioblastoma. IORT using the Xoft Axxent eBx System is no worse than (non-inferior) GliaSite radiation therapy when used as stand-alone radiation treatment immediately following maximal safe neurosurgical resection in patients with recurrent glioblastoma multiforme (GBM).

DETAILED DESCRIPTION:
Device Description: The Xoft Axxent Electronic Brachytherapy System is a device that delivers radiation at a high dose rate. It is designed for use with Axxent applicators to treat lesions, tumors, and conditions in or on the body where radiation is indicated. The Axxent System and Applicators are FDA cleared under 510(k)s K050843, K072683, K090914 and K122951.

The purpose of this trial is to assess the overall survival of patients treated with the Xoft Axxent eBx System for single-fraction IORT following maximal neurosurgical resection of recurrent glioblastoma. A historical comparison will be made for surgical excision and GliaSite radiation therapy (Chan 2005), which resulted in a median OS of 9.1 months.

Radiation is delivered to the target tissue (adjacent to the resection margins). It avoids treatment delays and eliminates weeks of post-surgical radiation therapy during which residual cancer cells might proliferate.

ELIGIBILITY:
Inclusion Criteria:

1. Potentially-resectable, histologically proven recurrent GBM
2. Subject must be ≥ 18 years of age
3. Subject must have a Karnofsky Performance Score ≥ 70%
4. Subject must have had a T1 weighted 3D MRI with Gadolinium enhancement within fourteen (14) days prior to surgery
5. Women of child-bearing potential must have a negative pregnancy test within one week of IORT treatment
6. Subjects of child-bearing potential must agree to use adequate contraceptive precautions and not to breastfeed (if applicable)

Exclusion Criteria:

1. More than three relapses
2. Subject has multi-centric disease
3. Subject has tumors in or near (less than 10mm from tumor margin) critical brain structures, that would exclude sufficient dose delivery to the tumor: such as:

   1. Optic Chiasm
   2. Optic Nerve
4. Women who are pregnant or nursing. Women with child-bearing potential or sexually active men that are not willing/able to use medically acceptable forms of contraception
5. Subject has contraindications for MRI with or without gadolinium injections
6. Subject has contraindications for anesthesia or surgery
7. Subject is on another therapeutic clinical trial concurrently
8. Subject had previous radiation for GBM less than 3 month earlier
9. Prior history of standard dose of Central Nervous System (CNS) of more than 60 Gy

Intra-Operative Exclusion Criteria

1. Frozen section does not show any sign of malignant tissue
2. Dose at any organ at risk will exceed 10 Gy including:

   1. Chiasm
   2. Optic Nerve

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-03-05 (Actual); Primary Completion 2023-11-03 (Actual); Study Completion 2023-11-03 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is Overall Survival (OS) | Overall Survival (OS) will be defined as the interval from enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to three years.
  The primary study goal is to assess Overall Survival (OS) of subjects treated with the Xoft Axxent Electronic Brachytherapy (eBx)® System when used for single-fraction, intra-operative radiation therapy (IORT) following maximal safe neurosurgical resection of recurrent glioblastoma for patients.
Patients treated with Xoft IORT device median overall survival (OS) | Overall Survival (OS) will be defined as the interval from enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to three years.
  The median and mean OS with Xoft will be calculated

SECONDARY OUTCOMES:
Local Progression-free Survival (PFS) | LocPFS will be assessed at baseline, Month 2, Month 6, then every 6 months until Year 3 follow-up.
  Local PFS will be assessed at following intra-operative treatment with the Xoft Axxent Electronic Brachytherapy System following maximal safe neurosurgical resection.
Quality of Life Assessment (Fact-Br) | QOL will be assessed at baseline, Month 2, Month 6, then every 6 months until Year 3 follow-up.
  To assess Quality of Life Status at baseline and following intra-operative treatment with the Xoft Axxent Electronic Brachytherapy System following maximal safe neurosurgical resection. The FACT-Br questionnaire assesses subjects on a scale of 0 (minimum) to 4 (maximum), 0 equal to "Not at all" and 4 equal to "Very Much"
Karnofsky Performance Status (KPS) | KPS will be assessed at baseline, Month 2, Month 6, then every 6 months until Year 3 follow-up.
  To assess Karnofsky Performance Status at baseline and following intra-operative treatment with the Xoft Axxent Electronic Brachytherapy System following maximal safe neurosurgical resection. The KPS grades from 100 to 0. 0, the lower score the worst the survival for the most serious illness. 100, the higher score, survival close to normal limits, no complaints.
Radiation-related Neurotoxicity | Radiation-related Neurotoxicity will be assessed at baseline, Month 2, Month 6, then every 6 months until Year 3 follow-up.
  Assess the rate of radiation-related neurotoxicity in subjects treated with the Xoft Axxent electronic Brachytherapy System when used for single-fraction, intra-operative radiation therapy treatment following maximal safe neurosurgical resection.
The rate and severity of Adverse Events (AEs), Adverse Device Effects (ADEs), and Unanticipated Adverse Device Effects (UADEs) | UADEs will be assessed at baseline, Month 2, Month 6, then every 6 months until Year 3 follow-up.
  The rate and severity of Adverse Events (AEs), Adverse Device Effects (ADEs), and Unanticipated Adverse Device Effects (UADEs) will be assessed at the time of treatment and at all follow-up visits. All Grade 3 or higher adverse events will be followed until resolution. Each event will be classified according to:
  * Device Related
  * Procedure Related
  * Radiation Related

CONTACTS AND LOCATIONS:
Overall Officials: David A Wiles, MD, Principal Investigator — Parkridge Medical Center - Neurosurgery
Locations (1):
- Parkridge Medical Center - Neurosurgery, Chattanooga, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wallner KE, Galicich JH, Krol G, Arbit E, Malkin MG. Patterns of failure following treatment for glioblastoma multiforme and anaplastic astrocytoma. Int J Radiat Oncol Biol Phys. 1989 Jun;16(6):1405-9. doi: 10.1016/0360-3016(89)90941-3. PMID 2542195
- [Background] Gaspar LE, Fisher BJ, Macdonald DR, LeBer DV, Halperin EC, Schold SC Jr, Cairncross JG. Supratentorial malignant glioma: patterns of recurrence and implications for external beam local treatment. Int J Radiat Oncol Biol Phys. 1992;24(1):55-7. doi: 10.1016/0360-3016(92)91021-e. PMID 1512163
- [Background] Choucair AK, Levin VA, Gutin PH, Davis RL, Silver P, Edwards MS, Wilson CB. Development of multiple lesions during radiation therapy and chemotherapy in patients with gliomas. J Neurosurg. 1986 Nov;65(5):654-8. doi: 10.3171/jns.1986.65.5.0654. PMID 3021931
- [Background] Mallick S, Benson R, Hakim A, Rath GK. Management of glioblastoma after recurrence: A changing paradigm. J Egypt Natl Canc Inst. 2016 Dec;28(4):199-210. doi: 10.1016/j.jnci.2016.07.001. Epub 2016 Jul 28. PMID 27476474
- [Background] Goryaynov SA, Gol'dberg MF, Golanov AV, Zolotova SV, Shishkina LV, Ryzhova MV, Pitskhelauri DI, Zhukov VY, Usachev DY, Belyaev AY, Kondrashov AV, Shurkhay VA, Potapov AA. [The phenomenon of long-term survival in glioblastoma patients. Part I: the role of clinical and demographic factors and an IDH1 mutation (R 132 H)]. Zh Vopr Neirokhir Im N N Burdenko. 2017;81(3):5-16. doi: 10.17116/neiro20178135-16. Russian. PMID 28665384
- [Background] Haj A, Doenitz C, Schebesch KM, Ehrensberger D, Hau P, Putnik K, Riemenschneider MJ, Wendl C, Gerken M, Pukrop T, Brawanski A, Proescholdt MA. Extent of Resection in Newly Diagnosed Glioblastoma: Impact of a Specialized Neuro-Oncology Care Center. Brain Sci. 2017 Dec 25;8(1):5. doi: 10.3390/brainsci8010005. PMID 29295569
- [Background] Hardesty DA, Sanai N. The value of glioma extent of resection in the modern neurosurgical era. Front Neurol. 2012 Oct 18;3:140. doi: 10.3389/fneur.2012.00140. eCollection 2012. PMID 23087667
- [Background] Krivoshapkin A, Sergeev G, Gaytan A, Kurbatov V, Kiselev R, Kalneus L. Effect of pre- and postoperative tumor volumetric parameters on the life expectancy of patients with brain glioblastomas. Bull Neurol Psychiatry Neurosurg. 2016;6:59-67.
- [Background] Krivoshapkin AL, Sergeev GS, Gaytan AS, Kurbatov VP, Kalneus LE, Tarantsev EG. New software for objective evaluation of brain glioblastoma resection degree. Zh Vopr Neirokhir Im N N Burdenko. 2014;78(5):33-9; discussion 40. English, Russian. PMID 25406906
- [Background] Louis DN, Perry A, Reifenberger G, von Deimling A, Figarella-Branger D, Cavenee WK, Ohgaki H, Wiestler OD, Kleihues P, Ellison DW. The 2016 World Health Organization Classification of Tumors of the Central Nervous System: a summary. Acta Neuropathol. 2016 Jun;131(6):803-20. doi: 10.1007/s00401-016-1545-1. Epub 2016 May 9. PMID 27157931
- [Background] Weller M, van den Bent M, Tonn JC, Stupp R, Preusser M, Cohen-Jonathan-Moyal E, Henriksson R, Le Rhun E, Balana C, Chinot O, Bendszus M, Reijneveld JC, Dhermain F, French P, Marosi C, Watts C, Oberg I, Pilkington G, Baumert BG, Taphoorn MJB, Hegi M, Westphal M, Reifenberger G, Soffietti R, Wick W; European Association for Neuro-Oncology (EANO) Task Force on Gliomas. European Association for Neuro-Oncology (EANO) guideline on the diagnosis and treatment of adult astrocytic and oligodendroglial gliomas. Lancet Oncol. 2017 Jun;18(6):e315-e329. doi: 10.1016/S1470-2045(17)30194-8. Epub 2017 May 5. PMID 28483413
- [Background] van Linde ME, Brahm CG, de Witt Hamer PC, Reijneveld JC, Bruynzeel AME, Vandertop WP, van de Ven PM, Wagemakers M, van der Weide HL, Enting RH, Walenkamp AME, Verheul HMW. Treatment outcome of patients with recurrent glioblastoma multiforme: a retrospective multicenter analysis. J Neurooncol. 2017 Oct;135(1):183-192. doi: 10.1007/s11060-017-2564-z. Epub 2017 Jul 20. PMID 28730289
- [Background] Ringel F, Pape H, Sabel M, Krex D, Bock HC, Misch M, Weyerbrock A, Westermaier T, Senft C, Schucht P, Meyer B, Simon M; SN1 study group. Clinical benefit from resection of recurrent glioblastomas: results of a multicenter study including 503 patients with recurrent glioblastomas undergoing surgical resection. Neuro Oncol. 2016 Jan;18(1):96-104. doi: 10.1093/neuonc/nov145. Epub 2015 Aug 4. PMID 26243790
- [Background] Landy HJ, Feun L, Schwade JG, Snodgrass S, Lu Y, Gutman F. Retreatment of intracranial gliomas. South Med J. 1994 Feb;87(2):211-4. doi: 10.1097/00007611-199402000-00013. PMID 8115886
- [Background] Ammirati M, Galicich JH, Arbit E, Liao Y. Reoperation in the treatment of recurrent intracranial malignant gliomas. Neurosurgery. 1987 Nov;21(5):607-14. doi: 10.1227/00006123-198711000-00001. PMID 2827051
- [Background] Harsh GR 4th, Levin VA, Gutin PH, Seager M, Silver P, Wilson CB. Reoperation for recurrent glioblastoma and anaplastic astrocytoma. Neurosurgery. 1987 Nov;21(5):615-21. doi: 10.1227/00006123-198711000-00002. PMID 2827052
- [Background] Pace A, Dirven L, Koekkoek JAF, Golla H, Fleming J, Ruda R, Marosi C, Le Rhun E, Grant R, Oliver K, Oberg I, Bulbeck HJ, Rooney AG, Henriksson R, Pasman HRW, Oberndorfer S, Weller M, Taphoorn MJB; European Association of Neuro-Oncology palliative care task force. European Association for Neuro-Oncology (EANO) guidelines for palliative care in adults with glioma. Lancet Oncol. 2017 Jun;18(6):e330-e340. doi: 10.1016/S1470-2045(17)30345-5. PMID 28593859
- [Background] Lederman G, Wronski M, Arbit E, Odaimi M, Wertheim S, Lombardi E, Wrzolek M. Treatment of recurrent glioblastoma multiforme using fractionated stereotactic radiosurgery and concurrent paclitaxel. Am J Clin Oncol. 2000 Apr;23(2):155-9. doi: 10.1097/00000421-200004000-00010. PMID 10776976
- [Background] Young B, Oldfield EH, Markesbery WR, Haack D, Tibbs PA, McCombs P, Chin HW, Maruyama Y, Meacham WF. Reoperation for glioblastoma. J Neurosurg. 1981 Dec;55(6):917-21. doi: 10.3171/jns.1981.55.6.0917. PMID 6271933
- [Background] Bloch O, Han SJ, Cha S, Sun MZ, Aghi MK, McDermott MW, Berger MS, Parsa AT. Impact of extent of resection for recurrent glioblastoma on overall survival: clinical article. J Neurosurg. 2012 Dec;117(6):1032-8. doi: 10.3171/2012.9.JNS12504. Epub 2012 Oct 5. PMID 23039151
- [Background] Ruben JD, Dally M, Bailey M, Smith R, McLean CA, Fedele P. Cerebral radiation necrosis: incidence, outcomes, and risk factors with emphasis on radiation parameters and chemotherapy. Int J Radiat Oncol Biol Phys. 2006 Jun 1;65(2):499-508. doi: 10.1016/j.ijrobp.2005.12.002. Epub 2006 Mar 6. PMID 16517093
- [Background] Miyatake S, Nonoguchi N, Furuse M, Yoritsune E, Miyata T, Kawabata S, Kuroiwa T. Pathophysiology, diagnosis, and treatment of radiation necrosis in the brain. Neurol Med Chir (Tokyo). 2015;55(1):50-9. doi: 10.2176/nmc.ra.2014-0188. Epub 2014 Dec 20. PMID 25744350
- [Background] Nguyen D, Rwigema JC, Yu VY, Kaprealian T, Kupelian P, Selch M, Lee P, Low DA, Sheng K. Feasibility of extreme dose escalation for glioblastoma multiforme using 4pi radiotherapy. Radiat Oncol. 2014 Nov 7;9:239. doi: 10.1186/s13014-014-0239-x. PMID 25377756
- [Background] Veldwijk MR, Zhang B, Wenz F, Herskind C. The biological effect of large single doses: a possible role for non-targeted effects in cell inactivation. PLoS One. 2014 Jan 22;9(1):e84991. doi: 10.1371/journal.pone.0084991. eCollection 2014. PMID 24465461
- [Background] Herskind C, Wenz F. Radiobiological aspects of intraoperative tumour-bed irradiation with low-energy X-rays (LEX-IORT). Transl Cancer Res. 2014;3(1):3-17. doi:10.3978/j.issn.2218-676X.2014.01.06.
- [Background] Bensaleh S, Bezak E, Borg M. Review of MammoSite brachytherapy: advantages, disadvantages and clinical outcomes. Acta Oncol. 2009;48(4):487-94. doi: 10.1080/02841860802537916. PMID 19031175
- [Background] Davis ME. Glioblastoma: Overview of Disease and Treatment. Clin J Oncol Nurs. 2016 Oct 1;20(5 Suppl):S2-8. doi: 10.1188/16.CJON.S1.2-8. PMID 27668386
- [Background] Martinez-Garcia M, Alvarez-Linera J, Carrato C, Ley L, Luque R, Maldonado X, Martinez-Aguillo M, Navarro LM, Vaz-Salgado MA, Gil-Gil M. SEOM clinical guidelines for diagnosis and treatment of glioblastoma (2017). Clin Transl Oncol. 2018 Jan;20(1):22-28. doi: 10.1007/s12094-017-1763-6. Epub 2017 Oct 30. PMID 29086250
- [Background] Stupp R, Tonn JC, Brada M, Pentheroudakis G; ESMO Guidelines Working Group. High-grade malignant glioma: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2010 May;21 Suppl 5:v190-3. doi: 10.1093/annonc/mdq187. No abstract available. PMID 20555079
- [Background] Scanderbeg DJ, Alksne JF, Lawson JD, Murphy KT. Novel use of the Contura for high dose rate cranial brachytherapy. Med Dosim. 2011 Winter;36(4):344-6. doi: 10.1016/j.meddos.2010.08.001. Epub 2010 Dec 8. PMID 21144735
- [Background] Zamzuri I, Rahman GI, Muzaimi M, Jafri AM, Nik Ruzman NI, Lutfi YA, Biswal BM, Nazaruddin HW, Mar W. Polymodal therapy for high grade gliomas: a case report of favourable outcomes following intraoperative radiation therapy. Med J Malaysia. 2012 Feb;67(1):121-2. PMID 22582564
- See also: Patterns of failure following treatment for glioblastoma multiforme and anaplastic astrocytoma — http://www.ncbi.nlm.nih.gov/pubmed/2542195
- See also: Supratentorial malignant glioma: patterns of recurrence and implications for external beam local treatment. — http://www.ncbi.nlm.nih.gov/pubmed/1512163
- See also: Development of multiple lesions during radiation therapy and chemotherapy in patients with gliomas — https://doi.org/10.3171/jns.1986.65.5.0654
- See also: Management of glioblastoma after recurrence: A changing paradigm. — http://doi.org/10.1016/j.jnci.2016.07.001
- See also: The Phenomenon of Long-Term Survival in Glioblastoma Patients. Part I: The Role of Clinical and Demographic Factors and an IDH1 Mutation — http://doi.org/10.17116/neiro20178135-16
- See also: The Value of Glioma Extent of Resection in the Modern Neurosurgical Era — https://www.frontiersin.org/article/10.3389/fneur.2012.00140
- See also: The 2016 World Health Organization Classification of Tumors of the Central Nervous System: a summary — http://doi.org/10.1007/s00401-016-1545-1
- See also: European Association for Neuro-Oncology (EANO) guideline on the diagnosis and treatment of adult astrocytic and oligodendroglial gliomas. — http://doi.org/10.1016/S1470-2045(17)30194-8
- See also: Treatment outcome of patients with recurrent glioblastoma multiforme: a retrospective multicenter analysis — http://doi.org/10.1007/s11060-017-2564-z
- See also: Retreatment of intracranial gliomas — http://www.ncbi.nlm.nih.gov/pubmed/8115886
- See also: Reoperation in the treatment of recurrent intracranial malignant gliomas. — http://www.ncbi.nlm.nih.gov/pubmed/2827051
- See also: Reoperation for recurrent glioblastoma and anaplastic astrocytoma. — http://www.ncbi.nlm.nih.gov/pubmed/2827052
- See also: Novel Use of the Contura for High Dose Rate Cranial Brachytherapy — http://doi.org/10.1016/j.meddos.2010.08.001
- See also: Polymodal therapy for high grade gliomas: a case report of favourable outcomes following intraoperative radiation therapy. — http://www.ncbi.nlm.nih.gov/pubmed/22582564.